CLINICAL TRIAL: NCT04554953
Title: A Multi-center, Prospective Observational Study to Evaluate the Effectiveness of a Combination Drug Including Fimasartan and Statins in Patients With Hypertension and Dyslipidemia
Brief Title: A Combination Drug Including Fimasartan and Statins in Patients With Hypertension and Dyslipidemia
Acronym: FIMASTAR
Status: Completed | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-FMS-OS-406
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Hypertension and Dyslipidemia
Keywords: Fimasartan and Statins
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Combination drug containing fimasartan and statins — Patients who correspond to one of the following:
  1. Patients who are planning to be treated with a combination drug containing fimasartan and statins after being newly diagnosed with essential hypertension and primary hypercholesterolemia
  2. Patients who are planning to switch to a combination drug of fimasartan and statins, among those who have been diagnosed with essential hypertension or primary hypercholesterolemia and are receiving hypertension treatment that is containing an ARB or dyslipidemia treatment that is containing a statin
  3. Patients who are planning to switch to a combination drug of fimasartan and statins, among those who have been diagnosed with essential hypertension and primary hypercholesterolemia and are receiving hypertension treatment that is containing an ARB and dyslipidemia treatment that is containing a statin

SUMMARY:
The primary objective of this study is to evaluate the effectiveness of a combination drug containing fimasartan and statins on the control of hypertension and dyslipidemia, and the secondary objective is to evaluate the drug cost reduction effect, patients' satisfaction level and safety of the combination drug administration.

DETAILED DESCRIPTION:
This study is designed as a non-interventional, multicenter, prospective observational study for patients with hypertension and dyslipidemia. If a patient voluntarily provides written consent to provide information for this study, the enrollment number will be assigned to subjects who meet the inclusion/exclusion criteria, and follow-up will be conducted for approximately 12 weeks. Pre-specified study-related data will be collected in the case report form during the observation period.

This is an observational study, and the number or interval of subjects' visits to the hospital is determined by the investigators' clinical judgment under actual medical circumstances in principle. Whether to participate in this study will not affect the patients' treatment (physician's prescription or diagnostic, therapeutic decisions).

The follow-up time points specified below indicate the time points of data collection. That is, the schedule of subjects' visits is freely determined by the investigators based on the medical condition of the subjects regardless of the follow-up time points specified in this protocol, but data that are generated during the study period and are deemed necessary in relation to the study may be collected in the case report form.

ELIGIBILITY:
Inclusion Criteria:

Participation in this study is possible only if all of the inclusion criteria below are satisfied.

1. Patients who provide written consent on the consent form for use of personal information after listening to explanations regarding the purpose, method, etc. of this study
2. Adult males and females aged 19 years or above
3. Patients who correspond to one of the following:

<!-- -->

1. Patients who are planning to be treated with a combination drug containing fimasartan and statins after being newly diagnosed with essential hypertension and primary hypercholesterolemia
2. Patients who are planning to switch to a combination drug of fimasartan and statins, among those who have been diagnosed with essential hypertension or primary hypercholesterolemia and are receiving hypertension treatment that is containing an ARB or dyslipidemia treatment that is containing a statin
3. Patients who are planning to switch to a combination drug of fimasartan and statins, among those who have been diagnosed with essential hypertension and primary hypercholesterolemia and are receiving hypertension treatment that is containing an ARB and dyslipidemia treatment that is containing a statin 4. The following test results available within 4 weeks prior to the enrollment date

   * Total Cholesterol (TC)

     * HDL-C ③ Triglyceride (TG) ④ LDL-C or LDL-C (Friedewald formula*)

       * non-HDL-C (Total cholesterol - HDL-C (mg/dL)) *LDL-C = Total cholesterol - HDL-C - (triglyceride/5) (mg/dL)

Exclusion Criteria:

Patients cannot participate in this study if any of the following exclusion criteria is applicable.

1. Contraindication according to the drug labeling of the combination drug ingredients (fimasartan, amlodipine) for hypertension containing fimasartan
2. Contraindication according to the drug labeling of statins (rosuvastatin, atorvastatin)
3. Secondary hypertension or suspected secondary hypertension - Aortic coarctation, hyperaldosteronemia, renal artery stenosis, renal hypertension, pheochromocytoma, Cushing's syndrome, polycystic kidney disease, etc.
4. Secondary dyslipidemia or suspected secondary dyslipidemia

   - Nephrotic syndrome, dysproteinemia, obstructive liver disease, Cushing's syndrome, etc.
5. Patients currently hospitalized or scheduled to be hospitalized
6. If an investigational drug has been administered within 12 weeks of the enrollment date, or if participation in another clinical study during this study participation period is planned
7. Patients who are deemed ineligible for study participation at the discretion of the investigators for other reasons

   -

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10,990 subjects This study involves patients with hypertension and dyslipidemia, and its purpose is to investigate the control rate of hypertension and dyslipidemia, drug cost reduction effect, patients' satisfaction level, and rare adverse events of combination drugs containing fimasartan and statins.
Sampling Method: Non-Probability Sample
Enrollment: 10877 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Blood pressure controlled to the target level | Week12
  Proportion of patients with blood pressure controlled to the target level (SiSBP, SiDBP) according to '2018 Guidelines for Management of Hypertension2' at Week 12. Site staff will be measuring Systolic and Diastolic Blood Pressure.
LDL-C controlled to the target level | Week 12
  Proportion of patients with LDL-C controlled to the target level according to 'Guidelines for Management of Dyslipidemia 4th Edition1' at Week 12

SECONDARY OUTCOMES:
Medication Satisfaction Questionnaire | Week 12
  Score (or change in the scores) of Medication Satisfaction Questionnaire (MSQ) assessed by patients at Week 12/ The scale title is MSQ(Medication satisfaction Questionnaire). The minimum score is '1' and maximum score is '7'. Higher score means a better outcome.
Average cost-effectiveness ratio (ACER) | Week 12
  Average cost-effectiveness ratio (ACER) of the study drug at Week 12
both blood pressure and LDL-C controlled | Week 12
  Proportion of patients with both blood pressure and LDL-C controlled to the target level simultaneously at Week 12
non-HDL-C controlled | Week 12
  Proportion of patients with non-HDL-C controlled to the target level at Week 12
Change in blood pressure | Week 12
  Change in blood pressure at Week 12 from baseline
Change in Lipid panel | Week 12
  Lipid panel at Week 12 from baseline
  * Percent change in TC
  * Percent change in HDL-C
  * Percent change in TG
  * Percent change in LDL-C
  * Percent change in non-HDL-C

CONTACTS AND LOCATIONS:
Locations (1):
- Chonnam National University Hospital, Gwangju, Jebong-ro, Jangseong-eup, Jangseong-gun, South Korea

IPD SHARING:
Plan to Share IPD: No